CLINICAL TRIAL: NCT03335618
Title: A First-in-Kind Randomized, Controlled Pilot Clinical Trial Testing Proactive vs Reactive Management of a Symptom Triad in Multiple Sclerosis
Brief Title: Coaching and Activity Tracking in Multiple Sclerosis - A Pilot Study
Acronym: CoachMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-20505
Record Dates: First submitted 2017-10-19; First posted 2017-11-08 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Multiple Sclerosis
Keywords: Activity; Mood
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Coaching and Monitoring (Experimental)
  Interventions: Other: Activity Monitoring and Symptom Coaching
- Passive Monitoring (Sham Comparator)
  Interventions: Other: Passive Activity Monitoring

INTERVENTIONS:
Other: Activity Monitoring and Symptom Coaching — Triggered check-ins by study personnel to keep participants on track to meet fitness goals
  Arms: Active Coaching and Monitoring
Other: Passive Activity Monitoring — Passive step tracking without check-ins
  Arms: Passive Monitoring

SUMMARY:
The purpose of this 12-week, exploratory pilot clinical trial is to continuously and remotely assess a triad of bothersome multiple sclerosis (MS) symptoms (BAM: bladder, ambulation, mood) and test the benefit of proactively treating these symptoms according to an evidence-based, multi-disciplinary, personalized protocol.

DETAILED DESCRIPTION:
MS is a chronic, debilitating disease of the central nervous system affecting approximately 2 million people worldwide and more than 400,000 individuals in the US. MS is the most common cause of non-traumatic neurological disability in young adults. Symptoms typically first afflict individuals during the prime of their professional and reproductive lives, between the ages of 20 and 40. Many affected individuals are unemployed, physically disabled, and at high risk for social isolation. While disease-modifying therapies (DMTs) can significantly reduce accumulation of disability in MS, patients still experience symptoms across a range of functional domains. Symptoms can include problems with bladder, walking, and mood (depression and anxiety). Often, these symptoms are only partially evaluated during routine MS clinic visits, and the long interval between clinic visits can result in them not being optimally managed.

The goal of the current study is to pilot a system of proactively monitoring a combination of symptoms (bladder, ambulation and mood) using an activity monitor and a smartphone.

Adult patients with MS who are experiencing symptoms in at least 2 of the 3 domains (bladder, ambulation, mood) will be enrolled. Visits will be at baseline (can be same day as routine visit to the MS clinic), and 3 months. Short surveys (<3 minutes to complete) will occur weekly, and longer surveys will occur at baseline, 6 weeks and 3 months. FitBit activity monitors will be worn for the entire 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Any individual above the age of 18 with a confirmed diagnosis of MS
* Access to a smartphone
* Access to Wi-Fi at home
* Able to walk (including with a cane or walker)
* Willing to fill out surveys at multiple time points

Exclusion Criteria:

* Clinician's assessment of cognitive, dexterity, or visual impairment limiting ability to use a smartphone and subsequent technologies required by the study
* Inability to walk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
Feasibility of an active symptom monitoring and intervention protocol | 12 weeks
  To evaluate feasibility of the intervention, we will calculate how many patients remain in the study, levels of patient satisfaction with the monitoring and intervention, and we will analyze patient and provider feedback.

SECONDARY OUTCOMES:
Improvement in ambulation symptoms in MS participants | 12 weeks
  Change in average daily step count according to FitBit step tracking. We will assess the mean observed change of daily steps between both the actively monitored group and the passively monitored group.
Improvement in mood symptoms in MS participants. | 12 weeks
  We will measure changes in the Center of Epidemiologic Studies Depression Scale-Revised (CES-D-R), which is a patient questionnaire that provides a measure of depression. It consists of 20 questions, each of which receives a score between 0 and 3, with higher scores indicating worse depression. The total CESD-R score (0-60) also permits categorization of no, mild, moderate and severe depression.
Improvement in bladder symptoms in MS participants. | 12 weeks
  At the end of the study, we will measure change in the Actionable Bladder Symptom Screening Tool (ABSST), which is a patient-reported scale that identifies patients who could benefit from lower urinary tract assessment and/or possibly treatment. It consists of 8 questions, each graded on 4 points, with higher scores indicating worse bladder function.

CONTACTS AND LOCATIONS:
Overall Officials: Riley M Bove, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bove R, Garcha P, Bevan C, et al. Towards a Tele-MSDS: an iterative method to assess the MS patient remotely. ECTRIMS. London 2016.
- [Background] Ritvo PG F, J. S., Miller, D. M., Andrews, H., Paty, D. W., LaRocca, N.G. . Multiple Sclerosis Quality of Life Inventory: A User's Manual. New York: National Multiple Sclerosis Society, 1997.
- [Background] Schwartz CE, Ayandeh A, Motl RW. Investigating the minimal important difference in ambulation in multiple sclerosis: a disconnect between performance-based and patient-reported outcomes? J Neurol Sci. 2014 Dec 15;347(1-2):268-74. doi: 10.1016/j.jns.2014.10.021. Epub 2014 Oct 18. PMID 25455299
- [Background] Motl RW, Pilutti L, Sandroff BM, Dlugonski D, Sosnoff JJ, Pula JH. Accelerometry as a measure of walking behavior in multiple sclerosis. Acta Neurol Scand. 2013 Jun;127(6):384-90. doi: 10.1111/ane.12036. Epub 2012 Dec 13. PMID 23240822
- [Background] Bove R, White CC, Giovannoni G, Glanz B, Golubchikov V, Hujol J, Jennings C, Langdon D, Lee M, Legedza A, Paskavitz J, Prasad S, Richert J, Robbins A, Roberts S, Weiner H, Ramachandran R, Botfield M, De Jager PL. Evaluating more naturalistic outcome measures: A 1-year smartphone study in multiple sclerosis. Neurol Neuroimmunol Neuroinflamm. 2015 Oct 15;2(6):e162. doi: 10.1212/NXI.0000000000000162. eCollection 2015 Dec. PMID 26516627
- [Background] Block VJ, Lizee A, Crabtree-Hartman E, Bevan CJ, Graves JS, Bove R, Green AJ, Nourbakhsh B, Tremblay M, Gourraud PA, Ng MY, Pletcher MJ, Olgin JE, Marcus GM, Allen DD, Cree BA, Gelfand JM. Continuous daily assessment of multiple sclerosis disability using remote step count monitoring. J Neurol. 2017 Feb;264(2):316-326. doi: 10.1007/s00415-016-8334-6. Epub 2016 Nov 28. PMID 27896433